CLINICAL TRIAL: NCT01949181
Title: Relationship Between Blood, Hair and Lung Metals/Metalloids Concentration (Cadmium, Iron, Copper, Nickel, Chrome, Arsenic, Vanadium, Beryllium, and Zinc) and Lung Cancer or Chronic Obstructive Pulmonary Disease.
Brief Title: Blood, Hair and Lung Concentrations of Metals and Metalloids in Patients With Lung Cancer or Chronic Obstructive Pulmonary Disease
Acronym: Métaux/Poumons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010/37
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Lung Cancer; Chronic Obstructive Pulmonary Disease; Emphysema; Lung Surgery
Keywords: Metals; Metalloids; Blood; Hair; Lung; Lung cancer; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Pulmonary Surgical Procedures

ARMS (1):
- Pulmonary cancer (Experimental)
  Interventions: Procedure: Lung surgery

INTERVENTIONS:
Procedure: Lung surgery

SUMMARY:
Prospective research to study the relationship between concentrations of metals/metalloids in blood, hair and lung tissue with the occurence of lung cancer or chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 to 75 years of age.
* Patients admitted for lung resection (either cancerous or non-cancerous) or lung transplant

Exclusion Criteria:

* Patients with mental or physical conditions that prevent them giving their agreement for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Metals/metalloids concentration | Blood, hair and lung tissue are sampled during lung surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Grassin Delyle, Study Chair — Hôpital Foch
Locations (2):
- France (2):
  - CHU de Poitiers, Chirurgie Cardiaque et Thoracique, Poitiers
  - Hopital Foch, Suresnes, Île-de-France Region